CLINICAL TRIAL: NCT03385044
Title: Comparison of Endotracheal Intracuff Pressure Between Two Cuff Sealing Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DongGuk University (Other)
Responsible Party: Principal Investigator, Junyong In, MD, PhD, Professor, DongGuk University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: J_In_2017-01
Record Dates: First submitted 2017-12-20; First posted 2017-12-28 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Endotracheal Tube
Keywords: Endotracheal tube; Intracuff pressure; Minimal occlusive volume technique; Spirometer; Endotracheal sealing

STUDY DESIGN:
Intervention Model Description: Two methods of cuff sealing will be applied in a random sequence to each patient.
Who Masked: Participant, Outcomes Assessor
Masking Description: The randomization table of a treatment sequence will be managed by the third person who will not involve in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cuff sealing by MOVT (Active Comparator): MOVT (minimal occlusive volume technique). The cuff sealing will be confirmed with MOVT, then the intracuff pressure will be measured.
  Interventions: Procedure: MOVT
- Cuff sealing by VE/VI ratio (Active Comparator): VE/VI ratio of Spirometer. The cuff sealing will be confirmed with VE/VI ratio of a spirometer, then the intracuff pressure will be measured.
  Interventions: Procedure: VE/VI ratio of Spirometer

INTERVENTIONS:
Procedure: MOVT — ETT cuff will be inflated till the disappearance of audible air leak on auscultation, while abdominal carbon dioxide (CO2) inflation is maintained with peak inspiratory pressure of 25 cm H2O during volume controlled ventilation. The patient will be in the Trendelenburg position.
  Arms: Cuff sealing by MOVT
Procedure: VE/VI ratio of Spirometer — ETT cuff will be inflated till the VE/VI ratio meets the initial VE/VI ratio, while abdominal CO2 inflation is maintained with peak inspiratory pressure of 25 cm H2O during volume controlled ventilation. The patient will be in the Trendelenburg position.
  Arms: Cuff sealing by VE/VI ratio

SUMMARY:
The endotracheal intracuff pressure is to be maintained at a low level to prevent trachea and nerve damages, and yet be high enough to secure air sealing. The objective of the study is to compare minimal occlusive volume technique (MOVT) and expired volume/inspired volume ratio (VE/VI ratio) from a spirometer method of endotracheal tube (ETT) cuff inflation with respect to the cuff pressure required to seal the airway during a laparoscopic surgery under general anesthesia. A study design is a randomized crossover trial in 35 patients. The primary outcome is the intracuff pressure of an endotracheal tube. The study consists of two cuff sealing methods separated by a period of 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status I, II
* Body mass index < 30 kg/m2
* Elective laparoscopic gynecologic surgery under general anesthesia in the Trendelenburg position

Exclusion Criteria:

* History of airway-related or pulmonary diseases/abnormalities
* When difficult intubation is anticipated
* History of general anesthesia within the past 3 months
* Pregnancy
* History of smoking

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2018-10-29 (Actual); Study Completion 2018-10-29 (Actual)

PRIMARY OUTCOMES:
Intracuff Pressure | From the start of cuff inflation to the airway sealing, an average of 2 minutes
  The intracuff pressure of endotracheal tube when cuff sealing is achieved.

SECONDARY OUTCOMES:
Intracuff air volume | From the start of cuff inflation to the airway sealing, an average of 2 minutes
  The intracuff air volume of endotracheal tube when cuff sealing is achieved.

CONTACTS AND LOCATIONS:
Overall Officials: Junyong In, MD, PhD, Principal Investigator — DongGuk University
Locations (1):
- Dept. of anesthesiology and pain medicine, Dongguk University Ilsan Hospital, Goyang, Gyeonggido, South Korea